CLINICAL TRIAL: NCT00667979
Title: A Pilot, Randomized, Double-Blind, Placebo-Controlled, Crossover Study Evaluating the Efficacy and Safety of Vardenafil Versus Placebo Administered 12, 18 and 24 Hours Prior to Initiation of Sexual Intercourse in Subjects With ED
Brief Title: Evaluating the Efficacy of Vardenafil in Subjects With Erectile Dysfunction (ED) Administered 12, 18 or 24 Hours Prior to Intercourse
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer Healthcare AG
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11586
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — 10mg and 20mg to be taken 12, 18, 24 hours prior to sexual intercourse
  Arms: Arm 1
Drug: Placebo — Matching placebo
  Arms: Arm 2

SUMMARY:
Erectile dysfunction (ED) is defined as the inability to achieve or maintain an erection sufficient for satisfactory sexual performance. However, there remains no prospectively obtained data on the maximal time of effectiveness of vardenafil. The goal of the current study was to determine if vardenafil will significantly increase the percentage of successful intercourse attempts from 12 to 24 hours following dosing. A total of three time points 12, 18, and 24 hours were assessed in this pilot study to better quantify the effect of vardenafil.

ELIGIBILITY:
Inclusion Criteria:

* Men >/= 18 years of age
* ED >/= 6 months
* Stable sexual relationship for > 6 months

Exclusion Criteria:

* Primary hypoactive sexual desire
* History of myocardial infarction, stroke or life-threatening arrhythmia within prior 6 month
* Nitrate therapy
* Other exclusion criteria apply according to the Summary of Product Characteristics

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 264 (Actual)
Dates: Start 2004-09; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Sexual encounter profile Question 3 | 6 weeks

SECONDARY OUTCOMES:
Safety and Tolerability | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer